CLINICAL TRIAL: NCT03509168
Title: Efficacy and Safety of Pre-operative Vaginal Misoprostol in Reduction of Intraoperative Blood Loss During Myomectomy. Amulticentre Single Blind Randomized Trial.
Brief Title: The Efficacy and Safety of Preoperative Misoprostol in Blood-loss Reduction During Myomectomy.
Acronym: MM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Principal Investigator, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: myomectomy trial
Record Dates: First submitted 2018-03-21; First posted 2018-04-26 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: multicenter-randomized single blind controlled trial with a (1:1) allocation ratio.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol Pfizer Brand arm (Active Comparator): participants receive a single dose of 400mcg vaginal misoprostol preoperatively (60minutes before) during open myomectomy
  Interventions: Drug: Misoprostol Pfizer Brand
- No misoprostol arm (Other): standard of care
  Interventions: Other: Non-insertion of Misoprostol Pfizer Brand

INTERVENTIONS:
Drug: Misoprostol Pfizer Brand — insertion of a preoperative single dose 400 micrograms of Misoprostol Pfizer Brand placed vaginally
  Other Names: cytotec
  Arms: Misoprostol Pfizer Brand arm
Other: Non-insertion of Misoprostol Pfizer Brand — participants in this arm will receive the standard of care which in our setting involves the use of either a tourniquet to control intraoperative blood loss especially if the fibroids are large or rarely, other interventions like oxytocin, tranexamic acid, vasopressin and occasionally not using either of the interventions.
  Arms: No misoprostol arm

SUMMARY:
Open myomectomy remains the principal treatment for symptomatic fibroids in sub-Saharan countries irrespective of fertility desires. This however has got to be balanced against potential risks such as profuse hemorrhage; blood loss at open myomectomy remains dreary with the use of various pharmacologic agents yielding inconclusive results. This trial is aimed at exploring the benefit of preoperative use of a readily available uterotonic, Misoprostol in reduction of intraoperative blood loss during open myomectomy with the Null hypothesis stating: there is no difference in mean blood loss during open myomectomy whether one preoperatively inserts a single dose of 400mcg vaginal misoprostol or not.

Alternate hypothesis: single dose 400mcg vaginal Misoprostol given 60 minutes preoperatively during open myomectomy reduces intra-operative blood loss by at least 20% as measured by surgical mops and suction.

Participants from two referral hospitals in Uganda with symptomatic fibroids and scheduled for open myomectomy will be recruited. 48 women that meet the inclusion criteria and have none of the exclusion criteria and provide signed informed consent will be enrolled. The screening will be done on the gynecological wards and patients will be randomized to either the control or interventional arm by means of sealed, sequentially numbered opaque envelopes containing computer-generated random numbers. Blinding will affect theatre team and patients. Primary (blood loss as estimated by surgical mops and suction) and secondary endpoints (e.g. postoperative drop in Hb) will be calculated. Data analysis: Data will be analyzed on an intention-to-treat basis. Analysis will be done using STATA software 14.0. This will include descriptive statistics for measures of central tendency and dispersion. Student t-test and Mann Whitney U test will be used for mean blood loss. Stratification for age, parity, complaints, total fibroid mass and usage of other intraoperative blood-loss techniques will be analyzed. categorical data to be analyzed by coefficients.

Results of this study are meant to better inform clinicians about the use of misoprostol for this role and possibly include it in the management protocols for open myomectomy in Sub-Saharan countries where burden of blood products is strained.

DETAILED DESCRIPTION:
Uterine fibroids are the commonest benign gynecological tumors in pre-menopausal women affecting over 80% of African women by age of 50. Myomas are clinically apparent in approximately 12 to 25% of reproductive age women and noted coincidentally on pathological examination in approximately 80% of surgically excised uteri. Fibroids; clinically apparent in up to one third of women in reproductive age, cause significant morbidity including prolonged or heavy menstrual bleeding, pelvic pressure or pain, dyspareunia and in other cases, reproductive dysfunction; all of which affect their quality of life. Although, the definitive mode of management is complete uterine removal (Hysterectomy), a significant fraction of patients prefer preserving their uterus irrespective of fertility desires. Myomectomy remains the mainstay of management for such patients. Open myomectomy, is a major surgical procedure associated with considerable morbidity with significant intraoperative hemorrhage. Fletcher in 1996 reported that 23% patients undergoing open myomectomy lost over 1000ml of blood. Another study of 91 women who underwent this procedure for uterine size greater than 16 weeks, the operative blood loss ranged between 50ml and 3000 ml. Other series reported transfusion rates between 18% and 24%. Surgical hemorrhage may result in anemia, hypovolemia, and coagulation abnormalities.

Despite the many advances in therapeutic options for uterine masses, open myomectomy poses the most efficacious mode of management in resource limited settings for symptomatic relief in women that wish to preserve their uteri. Laparoscopic myomectomy would offer a relatively more cosmetic and blood-sparing alternative but the high costs and the need for proficient personnel have left its advent in developing countries elusive.

Numerous strategies to reduce blood loss during abdominal myomectomy both mechanical and pharmacologic techniques have been tried but excessive hemorrhage during abdominal myomectomy remains a challenge to gynecologic surgeons.

Pre-operative prostaglandins, have offered a more reliable and realistic hope in resource-limited settings to lower intraoperative blood loss. It stimulates uterine contractions and this leads to occlusion of the vessels supplying blood to the leiomyomas. These strong myometrial contractions induced by misoprostol indirectly cause relative avascularity in the myoma and contributes to a reduction in bleeding. This subsequently may redistribute the blood from the diseased uterus back to the circulation, hence reducing operative blood loss during abdominal myomectomy. A few studies done have demonstrated safety and efficacy.

The complications and burden of this hemorrhage are even greater in resource-limited settings. In Mulago National Referral Hospital, Misoprostol has not been assimilated into the standard of care for reduction of intraoperative blood loss during open myomectomy. This study aims to assess the efficacy and safety of Misoprostol in such settings.

PROBLEM STATEMENT Uterine fibroids are major cause of gynaecological clinic attendance worldwide with approximately 20-30% of females affected. In Uganda, however, the burden of uterine fibroids across the whole country is not well documented. Unpublished Records from Mulago hospital, Uganda show that of the 2,088 patients that presented at the gynaecological outpatient clinic between September 2015 and September 2017, 525 (25.14%) had symptomatic fibroids. Additionally, gynaecological emergency records reveal that 210 of 16,121 (1.30.%) emergency patients presented with uterine fibroids within the same period. (Mulago Hospital records, 2017) .

Symptomatic women complain about abnormal uterine bleeding, dyspareunia cyclic pelvic pain, and Infertility. Among the women with uterine fibroids who presented to Mulago Hospital Gynecological department between September 2015 to August 2017, 64 / 525 (12.2%) underwent open myomectomy. The major contributor to this low myomectomy rate was lack of theatre space for all consenting patients with uterine fibroids. Other reasons included scarcity of blood products to book prior to this elective case.

A previous study in Nigeria found that post-myomectomy complications ranged from post operative pyrexia (13.5%), blood loss warranting blood transfusion (12.8%), postoperative anaemia (10.4%), wound infection (8.7%), vault infection (5.1%) and prolonged hospital stay (4.2%).Wound dehiscence (2.5%), vesicovaginal fistula (0.3%), ureteric (0.3%) and bladder injuries (0.6%) were other complications recorded. The postoperative complications also result in increased costs to the already strained health system. In particular the excessive blood loss(>1000ml) encountered in open myomectomy poses great challenges to the surgeons in the current use of tourniquets, preoperative Gonadotrophin-releasing hormone (GnRH) agonists,clamping of the bilateral uterine and /or ovarian arteries, injection of vasopressin into myometrium for hemostasis and scarce blood resources. In Mulago hospital, about 42 of 64 (65.6%) women who underwent open myomectomy in 2015/2017 received blood transfusions and 2 (3.0 %) underwent hysterectomies due to intractable intraoperative bleeding.

The burden imposed on a resource-limited health setting with the direly needed scarce blood products potentially brought by avoidable and feasible measures to reduce blood loss is imminent. The availability, affordability and minimal side effects of a potentially effective uterotonic, prostaglandin E1 analogue, Misoprostol offers prospect in resource-constrained settings. A few studies done show efficacy.

This study is therefore meant to feed the need for a safer and effective method of intraoperative blood loss control within limited resource settings. In addition it will also contribute to the body of knowledge on use of misoprostol that will guide formation of national and local health protocols and policies.

OBJECTIVES:

General objective To determine the efficacy and safety of pre-operative 400mcg vaginal Misoprostol in the reduction of intra-operative hemorrhage during open myomectomy.

Specific objectives

* To compare the efficacy of administration of preoperative 400μg vaginal Misoprostol in reduction of intraoperative blood loss versus its non-administration during open myomectomy.
* To determine the safety of using preoperative 400μg vaginal Misoprostol during open myomectomy.

METHODS

Study design:

A multicenter-randomized double blind controlled trial with a (1:1) allocation ratio

Study setting:

Mulago Referral Hospital (central Uganda) and Lacor hospital (northern Uganda). A review of theatre records for the complete three months of January, February and March 2017 in each of these hospitals was done to ascertain the average number of open myomectomies.

Mulago National Referral Hospital is situated in Kampala, 2 kilometres from the city centre and serves as Makerere University College of Health Sciences teaching hospital as well as a National referral hospital for Uganda. Mulago hospital had eight open myomectomies done between the start of January and end of March 2017.

St. Mary's Hospital Lacor is a referral private not-for-profit (PNFP) hospital situated 5km out of Gulu town and is a Gulu university teaching hospital. It has a 482-bed capacity and does an average of 467 major surgeries per month. Lacor Hospital managed to perform 36 open myomectomy cases within the stipulated months.

Study duration Duration of Subject Participation Participant accrual to last between 72 to 96 hours depending on the duration of postoperative care. This includes the enrolment or the preoperative day, the operation day and 48-72 hours follow up post-operatively.

Study Period

The duration of study period will be approximately 3 months:

Participants' recruitment: this will be ongoing throughout the study period and will only be halted before if any of the stopping rules are encountered. (Refer to stopping rules ahead)

Determination of sample size

TARGET POPULATION:

Women of reproductive age with symptomatic uterine fibroids

STUDY POPULATION:

Symptomatic participants with fibroids going for open myomectomy

SAMPLING PROCEDURE:

Consecutive sampling as participants with the said symptoms presenting to the respective health units will be enrolled as they come. Those admitted to the gynecology wards with symptomatic fibroids scheduled for open myomectomy and meet the inclusion criteria will be enrolled. Participants will be enrolled into the study by proportion proportional to the size sampling. Participants' pre-operative Hb and anesthetic review to be performed. The research assistant on site who will then get informed consent for enrollment into study will identify them. Participants will then be issued a brown envelop or kit initially randomized to either arm and either administered an Misoprostol tablet or not. Patients in the control arm get the usual care. The respective research assistant will ensure transportation to and from theatre.

SAMPLE SIZE ESTIMATION Sample size estimation for testing mean differences of intraoperative blood lost between the Misoprostol arm and the non intervention arm;-

Assumptions:

* Sample size estimation is based on hypothesis that blood loss intra-operatively during open myomectomy will be comparable between the intervention (400mcg Misoprostol) and the control arm.
* Assuming a type 1 error of 5%, power (type II error) of 80% and mean blood loss of 621mls in the placebo arm based on previous studies (Eugene J Kongnyuy & Wiysonge, 2014); and a 20% reduction in blood loss when misoprostol will be used; - N= [(1/q1 + 1/q2) S2(Zα + Zβ)^2] / [μ1 - μ2]^2

N = (1/0.5 + 1/0.5)(121)2(1.96 + 0.84)2

N = 21 participants in each arm. Considering 10% estimation of loss to follow up Adjusted sample size = 23 participants in each arm Total estimated sample size = 46 participants.

RANDOMIZATION Sequence generation and Randomization Participants will be randomly assigned to either control or experimental group with a 1:1 allocation as per a computer generated randomization schedule stratified by site using permuted blocks of random sizes. An independent statistician will be responsible for this generation.

Allocation concealment In order to protect the randomization code until a participant has irrevocably been enrolled into the trial, the trial assistants at both sites will receive codes from trial statistician for each study kit of trial medicines per participant enrollment. Only the manufacturer (who will not participate in participant enrollment) and trial statistician will have access to the linked data of the study kit serial numbers and randomization of the participants.

Implementation.

Permuted blocked randomization with two arms so as to ensure a balance of numbers in each group will be used. Block randomization to be achieved by a computer generated sequence operated by the statistician. The computer-generated list of interventions will consist of blocks containing 400mcg Misoprostol and others without Misoprostol. A block size of 6 will be used. This will be divided into smaller blocks of 4:2 and will be changed along the way to avoid predicting.

Random allocation to each block will be made and patients allocated as per the flow of the block sequence indicated so as to achieve allocation concealment. This will ensure even distribution in both arms of the study. Study assistants will submit the patient's identification to the principal investigator who will transfer them to the statistician to enter these against the intervention allocated thus keeping the randomization code unknown to the study assistant.

Blinding single blind randomized controlled trial. Blinding will both patients and the theatre team.

Prepackaged sample of Misoprostol in sequentially numbered brown envelopes will be availed to the study assistant and administered to the participants.

The treatment assignment kit will be concealed until the participant is enrolled into the study through sending of serialized kits with no (random assignment) revealing information to the onsite pharmacists. This will ensure that the person enrolling participants does not know in advance which trial arm the next person will get, thus shielding knowledge of forthcoming assignments.

INTERVENTION:

Description of interventional drug Misoprostol (Cytotec®: trade name of Pfizer) is formulated as a white hexagonal tablet. It is supplied as a blister pack. Each tablet contains 200-mcg Misoprostol.

Dosage regimen All participants who are eligible for enrollment and have given consent, will then be randomized to either Misoprostol or control arm.

In the intervention group, single dose vaginal 400mcg Misoprostol will be administered 60 minutes preoperatively and those in the control group will not receive any misoprostol. The individuals in the control arm of this study will be given the standard of care at each of the study sites which entails non administration of misoprostol.

Participant Withdrawal Criteria

A participant included in the study, will be withdrawn from scheduled treatment if any of the following criteria is observed:

* Severe adverse events (AEs) with severity grade > 3
* Serious adverse events (SAEs)
* At the request of the participant (withdrawal of consent)
* At the discretion of the principal investigator Participants who are withdrawn from the study will be replaced. Patients who have withdrawn due to non-compliance will be receiving the standard of care outside the trial framework. In case of AEs or SAEs, whenever possible, they will be followed up for safety assessments until the clinical problems have resolved. Reasons for their withdrawal will be fully documented in the case report form (CRF) Adverse Event Assessments A complete physical examination will be carried out on all participants recruited and will involve, a general and a systemic examination. Safety and tolerability of the trial procedure will be assessed based on clinical and laboratory assessments during follow up, according to NIH/NCI Common Terminology Criteria for Adverse Events version 4.0. (CTCAE 2010) Adverse events will be recorded during the study period. The information on the occurrence of all adverse events will be obtained by questioning plus results recorded at physical examination. All AEs will be recorded on the Adverse Event Form in the CRF/data collection tool with the following information: duration (start and end dates); severity grade (mild, moderate, severe); pattern, causality (relationship to the study drugs) and action(s) taken and, as relevant, the endpoint.

Intensity/Severity: classification according to the NIH/NCI CTCAE into grade 1 (mild), 2 (moderate), 3 (severe) and 4 (potential life-threatening).

The investigator will comment (in the respective section of the CRF) on any change compared to baselines that are considered as clinically relevant.

Expedited Reporting of Serious Adverse Event The investigator will report serious adverse events (SAEs) occurring or observed during the period of the study to the Data Safety and Monitoring Committee (DSMC). As soon as an SAE has been noted, the alert form must be sent by phone call (then, send via email) within 24 hours after the SAE has been noted, this will be followed by "Serious Adverse Event Report" form (copies included in the Investigator's File) within 5 working days. In case of incomplete information, the investigator has to provide follow-up information as soon as possible, again using the SAE report form. Information will include participants' details, participant study number, date of administration, participant hospital number, study drug taken, onset of event, type of adverse event, classification of adverse event, relationship to study agent, unexpectedness, and follow-up. The principal investigator will provide the SAE report to National Ethics Committee if required. All SAE will also be record in AE page of the data collection form or Case Report Form (CRF).

DATA MANAGEMENT AND ANALYSIS PLAN Data collection and entry Data will be collected using a pretested questionnaire that the study investigator and assistants completed. The research assistant will follow the participant to theatre and gather information on the details of the procedure as directed by the CRF. The assistant will follow through to estimate the blood lost. Completeness and accuracy of the data will be checked daily and organized before storage. The principal investigator will clean, compile, code, store and double-enter the data into a computer data base using Epidata, which will then be analyzed on an intention-to-treat basis using STATA Data Handling and Record Keeping All trial data will be recorded on the collection tools or CRF (appendix III). Only the investigators and authorized co-workers, according to the list of Authorized Signatory Form (ASF), are authorized to make entries on the CRFs. CRFs should be completed in English.

Completed data collection tools will be dated and signed by the investigator All clinical data will be entered into hospital sheet from where back-translation will be made into the collection tools. Original lab data will be attached in hospital file and only the results will be transferred into data collection tools. Data collection tools will be kept under lock and key.

After completion of the collection tools by the investigator, the clinical monitor will review for completeness and accuracy before sending them to the statistician. The data will be double entered into a database (Epi-data software version 3.1) where computer checks are used to identify selected protocol violations and data errors. Requests for clarifications or correction will be sent to the investigator, if necessary. Statistical analysis will be carried out after all enquiries have been done and data has been locked. ID number (randomization number) will be used.

ANALYSIS OF THE RESULTS Description of Statistical Methods Data Analysis will be done using STATA version 14.0 software.

Dependent variables All primary and secondary endpoints for efficacy will be summarized using descriptive statistics for measurements of central tendency (mean, median) and dispersion (standard deviation, range, 95% C.I. values) or frequency and percentage, where appropriate. The main analysis of efficacy parameters will be done using the intention-to-treat approach. The student's t-test or Mann Whitney U test will be used to assess for difference in mean blood loss. A 95% confidence interval will be used and the coefficients between the two groups for mean intraoperative blood loss, mean in the difference of pre- and post-operative hemoglobin levels, mean duration of operation and transfusion rates will be analyzed as a measure of association. Significance will be denoted with a p value of 0.05 or less.

Secondary endpoints for safety will be summarized descriptively. AEs will be summarized with descriptive measures by time point (mean, median and standard deviation, range or 95% C.I. values) and classifications according to the reference ranges. The main analysis for safety variables will be done using the intention-to-treat (ITT) approach. Comparison of categorical variables (incidence of adverse events) between the two treatment groups will be done using χ2 or Fisher exact test. A table summarizing adverse events and tolerability will be generated. The endpoints will then be compared using a log rank test to determine if differences were statistically significant.

Independent variables Stratification will be done to assess independent effects of participants' characteristics on the different endpoints. Risk estimates for multiple strata will be examined using Mantel Haenzel (MH) estimates of the RR.

Figures and tables to present will include: Baseline Characteristics, Effect of misoprostol and standard care on mean amount of intraoperative blood loss, mean difference in hemoglobin concentration and operation times and parameters to indicate drug safety.

Direct Access to Source Data/Documents The investigator will provide written agreement that the investigator/institution will permit clinical monitors, institutional review board (IRB) review, and regulatory inspection with direct access to source documents.

Quality Control/Quality Assurance This study will be conducted in accordance with "Good Clinical Practice" (GCP) and all applicable regulatory requirements, including the latest version of the Declaration of Helsinki (October 2013) The investigator will implement and maintain quality assurance and quality control systems with written Standard Operating Procedures (SOPs) to assure the trial is conducted and data are generated, recorded, and reported in compliance with the protocol, GCP, and the applicable regulatory requirements.

The trial team will consist of 5 research nurses, a principal investigator and 2 trial clinical monitors. The research nurses will poses at least a diploma course in nursing.

Prior to the start of the trial, the investigator will ensure that all research personnel have gone through training in accordance with GCP. They will have revisions of drug administration and infection control. There will be a post-test to evaluate competence of research personnel before they can be involved in the trial.

Prior to the enrollment of any participant at the site, the investigator will review the protocol and all trial related procedures, information of study drugs, procedures for obtaining informed consent, procedures for reporting adverse experiences and procedures for completing the data collection tools.

Standardized digital weighing scales calibrated to two decimal points in grams will be availed to each of the sites. These will be reset to zero prior to every reading. Pre-weighed disposable dry mops will be used for each case.

Clinical monitor on a regular basis will schedule site-monitoring visits. During these visits, information recorded in the collection tools will be verified against source documents for accuracy and completion. The clinical monitor will review the informed consent procedure, product accountability and storage, trial documents and trial progress. The clinical monitor will verify that the investigator follows the approved protocol or amendments (if any), she/he will observe trial procedures and will discuss any problems with the investigator. Monitoring visits will be recorded in the Monitoring Log at the investigator's site.

Source data verification (verification of data by comparing collection tools' entries with original laboratory reports and other participant records of the investigator): All data will be checked for each participant. These will include: participant identification, informed consent, selection criteria, drug administration, adverse events, primary and secondary effectiveness and safety parameters. The investigator will arrange for the retention of the Participant Identification List for at least 15 years after completion or discontinuation of the trial. The investigator is required to retain all participant files and source documents for 10 years.

DATA SAFETY The data will be stored onto two separate drives and flash discs that are to be kept in separate and secure places. A questionnaire pre-test will be carried out before the study formally commences to recruit study personnel. They will be trained on the use of the questionnaire, patient approach, blinding, intervention administration, as well as assessment and monitoring for treatment success and failures. The questionnaires will be re-examined by the researcher to avoid any mistakes that will have been overlooked by the research assistants, before data compilation.

DATA SAFETY MONITORING COMMITTEE AND SAFETY MONITORING Data Safety and Monitoring Committee (DSMC) Members of Data Safety Monitoring Board (DSMB) will be composed of five members consisting of independent clinical experts. No investigator directly involved in the care of the subjects recruited will be a member of the DSMC. Ad hoc meetings can be convened if necessary. The principal investigator will be responsible for continuous close monitoring of all adverse effects that might occur on recruited subjects.

Participant Data Protection and Confidentiality The investigator and other members of the study team will keep confidential any information related to this study and all data and records generated in the course of conducting the study, and will not use the information, data, or records for any purpose other than those specified in this study.

Data collection tools or other documents will identify a patient by initials and number only. The investigator will keep in his file a Patient Identification List and Screening/Enrollment Log. At all times records will be referred to by code and not by name.

Interim analyses will be done once (at the midpoint of participant recruitment) during the trial to assess recruitment and safety of the participants on the study.The interim analysis will be done by an independent statistician on the DSMC and will consider the following stopping rules.

STOPPING RULES Pocock's approach of stopping rules will be used as it offers the same significance level at the interim analysis and final trial trial data analysis. This study will be halted if; -

1. Standards of care in the control of bleeding during open myomectomy change to involve preoperative misoprostol use prior to completion and publishing of the research results.
2. Mean difference in blood loss between the placebo arm and intervention arm is more than 30 % at interim analysis.
3. Lethality from intervention. Evidence of death of any participant from usage of vaginal misoprostol will culminate into immediate halt of the study.

ETHICAL CONSIDERATIONS:

Permission from regulatory/supervising bodies will be sought.

Confidentiality assurances The information provided by the patients will remain confidential. Nobody except principal investigator will have access to it. A study number known to the patient and the study personnel will be used instead of the name.

No Conflicts of Interest to declare.

Participant Information and Informed Consent All potential participants will be provided information regarding the study and allowed to make decisions of whether to participate or not with assurances of no compromise in care provided. Research assistants who will not be part of the care team will be involved in this screening of participants to minimize biases in recruitment

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age (15-49 years)
* Documented symptomatic uterine fibroids by ultrasound imaging
* Presenting to any of the selected hospitals within the study period.
* Scheduled for open myomectomy
* Willing to give informed consent

Exclusion Criteria:

* Previous uterine surgeries.
* Poorly controlled hypertension or diabetes
* History of a bleeding disorder, concurrent anticoagulant therapy, family history of bleeding disorder, prior history of deep venous thrombosis.
* Pregnancy
* Hemoglobin less than 10.5 g/dL at the time of surgery
* Prior treatment using GnRH analogues
* Intra-operative exclusion; pelvic endometriosis, adenomyosis, pelvic abcesses, pelvic malignancies

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-06-03 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss during open myomectomy in milliliters | immediate post-operative
  Soaked mops will be weighed and blood loss estimated by subtracting the soaked weight from the dry weight and by multiplying this by 1.060 (average density of human blood is 1.06g/ml); a volume in ml would be acquired. Only mops are intended to be routinely used during the operation for cleaning and clearing the operation field although measurement of blood collected in the suction cylinder in milliliters if used will also be added. Adequate mops will be provided to avoid any spillage onto the operating table polythene sheet. A standardized digital weighing scale will be availed in each operating room. Any spillage onto the bed, however, will be collected in a polythene sheet and poured into a measuring cylinder for quantification.

SECONDARY OUTCOMES:
duration of surgery | immediate postoperative
  from incision time to time for insertion of last stitch
duration of hospital stay | 4th postoperative day. (96 hours)
  number of days spent within the hospital post-operatively
need for blood transfusion | during and within 72 hours after open myomectomy
  hemodynamic instability during and after open myomectomy following profuse hemorrhage as assessed by the clinicians.
Serious adverse outcomes | 72 hours following open myomectomy
  death, massive transfusion >5 units of blood, development of deep venous thrombosis pulmonary edema and pulmonary embolism
drop in postoperative hemoglobin concentration | hemoglobin estimation done approximately 72 hours post-operatively
  Hemoglobin estimation done both pre- and post-operatively; difference between the two values to be a measure of amount of blood lost. patients that receive blood transfusion to be excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Moses Mugisha, Principal Investigator — Makerere University; Josephat Byamugisha, Professor, Study Chair — Makerere University
Locations (1):
- Makerere University, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: No